CLINICAL TRIAL: NCT04262947
Title: The Efficacy of Near-Infrared Vein Imaging for the Success of Placing Peripheral Venous Catheters in Adults With Difficult Venous Access
Brief Title: Efficacy of Near-Infrared Vein Imaging for Difficult IV Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID epidemic
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 20193166; NCT05051020 (obsolete NCT alias)
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-01

CONDITIONS: Catheterization, Peripheral
Keywords: Near-Infrared Vein Imaging; Difficult Venous Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Conventional Method (Active Comparator): Placement of peripheral venous catheter using conventional methods
  Interventions: Other: Conventional IV placement
- VeinViewer Visualization Only (Experimental): Use of a VeinViewer to visualize the most suitable target. Once the target has been identified and marked, the device will be placed aside and the peripheral venous catheter will be placed using conventional methods
  Interventions: Device: Near Infrared Vein Imaging; Other: Conventional IV placement
- Constant Imaging with VeinViewer (Experimental): Identification of the most suitable target and placement of a peripheral venous catheter under constant imaging with a VeinViewer
  Interventions: Device: Near Infrared Vein Imaging

INTERVENTIONS:
Device: Near Infrared Vein Imaging — Use of NI vein imaging device for visualization of veins during peripheral IV placement
  Other Names: VeinViewer Flex
  Arms: Constant Imaging with VeinViewer; VeinViewer Visualization Only
Other: Conventional IV placement — IV placement utilizing conventional methods
  Arms: Conventional Method; VeinViewer Visualization Only

SUMMARY:
The objective of this project is to define the effectiveness and therefore the role of NIR vein finders in adult patients with difficult peripheral venous access. The specific objective of the proposed randomized controlled trial is to test the clinical success rate of placing peripheral venous catheters in 'difficult' access patients using traditional peripheral venous catheter placement compared to two established methods utilizing NIR vein imaging. The investigators hypothesize that the capability to successfully place lasting peripheral venous catheters is increased with the adjunct of the imaging technology, reducing the number of failed needle sticks, reducing the number of peripheral venous catheters placed throughout a patient's hospital stay, and reducing the need for more invasive catheters such as PICC lines.

DETAILED DESCRIPTION:
The efficacy of NIR vein finders beyond the first line approach, particularly in patients that have failed conventional peripheral venous access methods or in patients that are expected to be a "difficult stick", is not established. Conflicting results have been reported in the pediatric literature regarding the subjective benefit of NIR light devices in patients with perceived difficult peripheral intravenous access. In addition, knowledge about the efficacy of these devices in the adult inpatient setting is mostly unknown. The aim of the present study is to address these knowledge gaps.

ELIGIBILITY:
Inclusion Criteria:

* non-pediatric in-hospital patients (≥15 years of age, inpatient and outpatient setting)
* willing to provide research authorization
* scheduled and consented to undergo peripheral venous cannulation of one of the upper extremities to be performed by one of the members of the Vascular Access Team
* determined to be a difficult peripheral venous access defined by one of the following criteria in alignment to the A-DIVA scale to be assessed by one of the members of the Vascular Access Team [8]:
* failed inspection for more than one visible or palpable suitable vein through conventional methods
* failed at least one attempt of peripheral venous cannulation through any methods
* history of difficult peripheral venous access
* greatest diameter of target vein less than 3mm determined by conventional methods

Exclusion Criteria:

* clinical contraindication for placement of peripheral venous catheter, including:
* severe bilateral upper extremity edema
* severe bilateral upper extremity skin burn
* severe bilateral upper extremity cellulitis
* history of bilateral axillary lymphadenectomy
* known severe cardiovascular or pulmonary compromise demanding minimization of procedure time, such as:
* severe shock with severe cardiovascular instability
* active CPR
* major uncontrolled hemorrhage
* any condition for which the primary healthcare provider is requesting emergent venous access
* scheduled PICC or midline catheter placement
* non-English-speaking patients if an interpreter is not available
* prisoner and any individual involuntarily confined or detained in a penal institution
* impaired capacity to make informed medical decisions

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schnelldorfer, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith AM, Mancini MC, Nie S. Bioimaging: second window for in vivo imaging. Nat Nanotechnol. 2009 Nov;4(11):710-1. doi: 10.1038/nnano.2009.326. PMID 19898521
- [Background] Kim JG, Xia M, Liu H. Extinction coefficients of hemoglobin for near-infrared spectroscopy of tissue. IEEE Eng Med Biol Mag. 2005 Mar-Apr;24(2):118-21. doi: 10.1109/memb.2005.1411359. No abstract available. PMID 15825855
- [Background] Chiao FB, Resta-Flarer F, Lesser J, Ng J, Ganz A, Pino-Luey D, Bennett H, Perkins C Jr, Witek B. Vein visualization: patient characteristic factors and efficacy of a new infrared vein finder technology. Br J Anaesth. 2013 Jun;110(6):966-71. doi: 10.1093/bja/aet003. Epub 2013 Feb 5. PMID 23384732
- [Background] Guillon P, Makhloufi M, Baillie S, Roucoulet C, Dolimier E, Masquelier AM. Prospective evaluation of venous access difficulty and a near-infrared vein visualizer at four French haemophilia treatment centres. Haemophilia. 2015 Jan;21(1):21-6. doi: 10.1111/hae.12513. Epub 2014 Oct 21. PMID 25335191
- [Background] Park JM, Kim MJ, Yim HW, Lee WC, Jeong H, Kim NJ. Utility of near-infrared light devices for pediatric peripheral intravenous cannulation: a systematic review and meta-analysis. Eur J Pediatr. 2016 Dec;175(12):1975-1988. doi: 10.1007/s00431-016-2796-5. Epub 2016 Oct 26. PMID 27785562
- [Background] Heinrichs J, Fritze Z, Klassen T, Curtis S. A systematic review and meta-analysis of new interventions for peripheral intravenous cannulation of children. Pediatr Emerg Care. 2013 Jul;29(7):858-66. doi: 10.1097/PEC.0b013e3182999bcd. PMID 23823270
- [Background] Johr M, Berger TM. Venous access in children: state of the art. Curr Opin Anaesthesiol. 2015 Jun;28(3):314-20. doi: 10.1097/ACO.0000000000000181. PMID 25827277
- [Background] Loon FHJV, Puijn LAPM, Houterman S, Bouwman ARA. Development of the A-DIVA Scale: A Clinical Predictive Scale to Identify Difficult Intravenous Access in Adult Patients Based on Clinical Observations. Medicine (Baltimore). 2016 Apr;95(16):e3428. doi: 10.1097/MD.0000000000003428. PMID 27100437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Method | VeinViewer Visualization Only | Constant Imaging With VeinViewer
Started | 13 | 13 | 12
Completed | 13 | 13 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Method | VeinViewer Visualization Only | Constant Imaging With VeinViewer | Total
Number analyzed (Participants) | 13 | 13 | 12 | 38
Age, Categorical [Count of Participants; unit: Participants] — Population: 38 patients is total number of study population
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 10 | 9 | 8 | 27
    >=65 years | 3 | 4 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 7 | 23
  Male | 4 | 6 | 5 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Initial IV Placement
Description: Rate of successful initial placement of a peripheral venous catheter (investigators have up to 30 minutes or ONE attempt before the study allows for change of technique to the preference of the Vascular Access Team member)
Time Frame: up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Method | VeinViewer Visualization Only | Constant Imaging With VeinViewer
Number analyzed (Participants) | 13 | 13 | 12
Participants | 10 | 6 | 6

ADVERSE EVENTS:
Time Frame: During hospital stay, an average of 4 days
Arm/Group | Conventional Method | VeinViewer Visualization Only | Constant Imaging With VeinViewer
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04262947/Prot_SAP_000.pdf